CLINICAL TRIAL: NCT01869153
Title: Monitoring Growth of Preterm Infants
Status: Terminated | Type: Observational
Why Stopped: Study expired; PI failed to submit study to IRB for continuing review
Sponsor: University of California, Davis (Other)
Responsible Party: Sponsor
Other Study IDs: 308519; UCD-308519 (Other: UCDavis)
Record Dates: First submitted 2013-05-27; First posted 2013-06-05 (Estimated); Last update posted 2018-09-20 (Actual); Status verified 2018-09

CONDITIONS: Prematurity
Keywords: Growth, weight
MeSH Terms: conditions — Premature Birth; Body Weight

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Preterm infants: Preterm infants born at either <32 weeks gestation or < 1750g birth weight

SUMMARY:
Growth is poor in preterm infants, partly due to difficulty identifying when growth is slow. The investigators will examine the use of a computer program to try and identify periods of growth slowing in preterm babies, and compare those results to the usual assessments made on patient care rounds.

DETAILED DESCRIPTION:
We wish to examine the use of a mathematical modeling system to see if it can detect poor growth better (and more quickly) than we can clinically. To do this, we need to know what the clinical team think about a baby's growth day-to-day. However, after rounds the fellow or NNP with fill in a sheet to say what the team thought about the baby's growth (was it okay, too slow, too fast etc.), and whether any changes were made to improve the baby's growth (e.g. increased feed volume, change in composition of feeds etc.). After the baby is discharged home, weight data from the EMR will be entered into the program to try and identify times where growth slowed (or where growth was faster than expected). We will compare the results of the computer program and the record of the clinical teams thoughts on the ward round, to see if the computer program identified growth slowing more quickly than the clinical team did.

ELIGIBILITY:
Inclusion Criteria:

1. Birth weight < 1750g gestational age < 32w at birth

   Exclusion Criteria:
2. Currently receiving parenteral nutrition or intravenous lipids

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Preterm infants of gestational age < 32w at birth, or <1750 weight at birth.
Sampling Method: Non-Probability Sample
Enrollment: 48 (Actual)
Dates: Start 2013-05; Primary Completion 2015-06-22 (Actual); Study Completion 2018-07-10 (Actual)

PRIMARY OUTCOMES:
Identification of growth slowing | Between birth and hospital discharge, an average of 10weeks
  At time of hospital discharge retrospectively collected data on daily weights (from the EMR) will be entered in to a computer program, to identify times where weight gain slowed significantly. This will be compared to the clinical assessment of the baby's growth made at the time (and recorded prospectively)

CONTACTS AND LOCATIONS:
Overall Officials: Ian Griffin, MD, Principal Investigator — University of California, Davis
Locations (1):
- NICU, University of California, Davis, Sacramento, California, United States